CLINICAL TRIAL: NCT05307744
Title: Effects of Lactobacillus Plantarum PS128 in Children With Autism Spectrum Disorder
Brief Title: Effects of Lactobacillus Plantarum PS128 in Children With ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Bened Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 202101416A3
Record Dates: First submitted 2022-03-14; First posted 2022-04-01 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PS128 (Experimental): Subjects will take PS128 capsules every day (2 capsules/day, once) for 12 weeks.
  Interventions: Dietary Supplement: PS128
- Placebo (Placebo Comparator): Subjects will take placebo capsules every day (2 capsules/day, once) for 12 weeks.
  Interventions: Other: Placebo
- Normal control (No Intervention): Normal control group are enrolled by invitation from the age and gender matched healthy children.

INTERVENTIONS:
Dietary Supplement: PS128 — Each PS128 capsule contained >3 × 10^10 colony forming units (CFU) with microcrystalline cellulose and weights 425 ± 25 mg.
  Arms: PS128
Other: Placebo — The placebo capsules only contained 425 ± 25 mg microcrystalline cellulose.
  Arms: Placebo

SUMMARY:
Autism spectrum disorder (ASD) is a neurodevelopmental disorder that can cause significant social, communication and behavioral deficits. Probiotics are regarded as active microorganisms. With sufficient amounts, probiotics can regulate intestinal flora, intestinal permeability, inflammation and antioxidant reactions in the body. These reactions may further promote health, regulate metabolic disease progression and prevent complications. Lactobacillus plantarum PS128 (PS128) was reported to be a psychobiotic in several animal and human studies which modulated the levels of neurotransmitters in different brain areas. This study is to evaluate whether the consumption of PS128 can improve the symptoms of patients with ASD. The current randomized, placebo-controlled trial was conducted to investigate the psychophysiological effects of PS128 in school children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age 7 to 12 years old.
* (2) PS128 group and placebo group: Children with autism spectrum disorder, confirmed by Autism Diagnostic Observation Schedule.
* (3) Normal control group: Children without autism spectrum disorder.

Exclusion Criteria:

* (1) Receiving antibiotics within one month.
* (2) Probiotics used in powder, capsule, or tablet in two weeks (except for Yogurt, Yogurt, Yakult and other related foods).
* (3) Patients with hepatobiliary gastrointestinal tract who have undergone surgery (except for hernia surgery and appendectomy)
* (4) Those with special diets (gluten-free, casein-free, high-protein, and ketogenic diet).
* (5) Those with a history of cancer.
* (6) Those who are allergic to lactic acid bacteria.
* (7) Not eligible judged by PI

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of total scores of Social Responsiveness Scale | Baseline, Week 12 and Week 16
  Social Responsiveness Scale can measure the autism clinical severity with the range from 65-260. The lower scores stand for better social responsiveness.

SECONDARY OUTCOMES:
Changes of total scores of Repetitive Behavior Scale-Revised | Baseline, Week 12 and Week 16
  Repetitive Behavior Scale-Revised is a questionnaire that focuses on repetitive behavior. The score ranges from 0-129. The lower scores stand for lower repetitive behavior.
Changes of total scores of Child Behavior Checklist | Baseline, Week 12 and Week 16
  Child Behavior Checklist is a parents' report questionnaire for behavioral and emotional problems. The lower scores stand for better behavioral and emotional regulation.
Changes of total scores of Adaptive Behavior Assessment System | Baseline, week 12 and Week 16W
  Adaptive Behavior Assessment System is a parents' report questionnaire for adaptive behavior. The score ranges from 9-171. The higher scores stand for better adaptive behavior.
Changes in accuracy of Frith-Happe animation | Baseline, Week 12 and Week 16
  A quick and objective test of Theory of Mind. 8 questions in total, the more correct questions stand for better Social Cognition.
Changes in accuracy of Eyes task | Baseline, Week 12 and Week 16
  An advanced test for Theory of Mind. 43 questions in total, the more correct questions stand for better social skills.
Changes of total scores of Aberrant Behavior Checklist | Baseline, Week 12 and Week 16
  Aberrant Behavior Checklist is a parents' report questionnaire for aberrant behavior. The lower scores stand for less aberrant behavior.
Visual Analogue Scale for GI symptoms | Baseline, week 12 and Week 16
  Visual Analogue Scale for GI symptoms was designed to measure the response of symptoms and well-being in patients after taking PS128. The score ranges from 0-10. The lower scores stand for less GI symptoms.
Changes of total scores of Emotional Dysregulation Inventory | Baseline, Week 12 and Week 16
  Emotional Dysregulation Inventory is a parents' report questionnaire for emotional dysregulation. The score ranges from 0-120. The lower scores stand for better emotional regulation.
Changes of total scores of Parenting Stress Index, Fourth Editon | Baseline, Week 12 and Week 16
  Parenting Stress Index is a parents' report questionnaire for parenting stress. The lower scores stand for lower parenting stress.
Assessment of Clinical Global Impression-Severity of Illness | Baseline, Week 12 and Week 16
  The Clinical Global Impression (CGI) is a clinician rated measure of illness severity, improvement, and efficacy of treatment. The CGI-I is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention.CGI Improvement scale: 1=very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; 7=Very much worse.
Assessment of Patient Global Impression of Change | Week 12 and Week 16
  The self-report measure Patient Global Impression of Change (PGIC) reflects a patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Gut microbiota | Baseline and Week 12
  Collect the DNA of fecal flora to test the diversity and abundance of gut microbiota as well as short chain fatty acids in Stool samples. The 16S rRNA gene amplicons will be prepared following the Illumina protocol for preparing the 16S metagenomic sequencing library.
MRI T1 | Baseline and Week 12
  Brain structural volumes (cm²)
functional MRI (resting-state/biological motion task) - BOLD signal | Baseline and Week 12
  Blood-oxygen-level-dependent (BOLD) signal is a measurement used in fMRI, which reflects the neural activity.
Diffusion Tensor Imaging (DTI) - FA | Baseline and Week 12
  Fractional anisotropy (FA) is a measurement used in DTI, which reflects the movement of water molecules. FA ranges from 0 to 1, the higher FA value may represent more intact axons.
Safety assessment - Albumin | Baseline and Week 12
  Safety is assessed function of liver and kidney such as albumin (6.6-8.7 g/dl).
Safety assessment - Total Protein | Baseline and Week 12
  Safety is assessed function of liver and kidney such as total protein (3.8-5.3 g/dl).
Safety assessment - ALP | Baseline and Week 12
  Safety is assessed function of liver and kidney such as ALP (40-129 IU/L).
Safety assessment - Total Bilirubin | Baseline and Week 12
  Safety is assessed function of liver and kidney such as total bilirubin (0.2-1.2 mg/dl).
Safety assessment - T-Cholesterol | Baseline and Week 12
  Safety is assessed function of liver and kidney such as T-Cholesterol (<170 mg/dL).
Safety assessment - Uric Acid | Baseline and Week 12
  Safety is assessed function of liver and kidney such as uric acid (3.4-7.6 mg/dl).
Safety assessment - BUN | Baseline and Week 12
  Safety is assessed function of liver and kidney such as BUN (6-20 mg/dl).
Safety assessment - Creatinine | Baseline and Week 12
  Safety is assessed function of liver and kidney such as creatinine (0.6-1.3 mg/dl).
Safety assessment - AST | Baseline and Week 12
  Safety is assessed function of liver and kidney such as AST (8-38 IU/L).
Safety assessment - ALT | Baseline and Week 12
  Safety is assessed function of liver and kidney such as ALT (4-44 IU/L).
Change in levels of exploratory blood-based biomarkers for inflammatory changes - MPO | Baseline and Week 12
  Inflammatory is assessed via a composite measure of circulating cytokines - MPO (ng/mL)
Change in levels of exploratory blood-based biomarkers for inflammatory changes - IL-1β | Baseline and Week 12
  Inflammatory is assessed via a composite measure of circulating cytokines - IL-1β (pg/mL)
Change in levels of exploratory blood-based biomarkers for inflammatory changes - TGF-β1 | Baseline and Week 12
  Inflammatory is assessed via a composite measure of circulating cytokines - TGF-β1 (pg/mL)
Change in levels of exploratory blood-based biomarkers for inflammatory changes - Eotaxin | Baseline and Week 12
  Inflammatory is assessed via a composite measure of circulating cytokines - Eotaxin (pg/mL)
Change in levels of exploratory blood-based biomarkers for inflammatory changes - IL-6 | Baseline and Week 12
  Inflammatory is assessed via a composite measure of circulating cytokines - IL-6 (ng/mL)
Change in levels of exploratory blood-based biomarkers for oxidative stress changes - Serotonin | Baseline and Week 12
  Oxidative stress is assessed via Serotonin (ng/mL).
Change in levels of exploratory blood-based biomarkers for oxidative stress changes - GABA | Baseline and Week 12
  Oxidative stress is assessed via GABA (umol/L).
Change in levels of exploratory blood-based biomarkers for oxidative stress changes - Cortisol | Baseline and Week 12
  Oxidative stress is assessed via Cortisol (nmol/L).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan